CLINICAL TRIAL: NCT03157440
Title: Validation of a Novel Device for Screening Patients With Symptoms of OSA
Brief Title: Novel Device for Screening Patients With Symptoms of OSA
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, To Kin Wang, Doctor, Chinese University of Hong Kong
Other Study IDs: 2016.661
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Sleep Apnea Syndromes
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ring oxymetry — a new type oxymetry wear on index finger like a ring

SUMMARY:
An innovative ring type oxymetry will be wore by patient undergoing sleep study to validate it's accuracy and usefulness as a screening device for patients with symptoms of OSA

ELIGIBILITY:
Inclusion Criteria:

* Patients above 18 years old and below 70 years old, both men and women

Exclusion Criteria:

* Patients requiring oxygen therapy or noninvasive ventilation;
* Patients with a diagnosis of chronic obstructive pulmonary disease, chronic heart failure, neuromuscular disease, insomnia, clinical symptoms of parasomnia, periodic limb movement, or narcolepsy.
* Patients on medication known to interfere with heart rate, such as beta-blockers, digoxin or calcium receptor antagonists.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with symptoms of OSA who will be undergoing sleep study for establishing a diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
the concordance of the ring oximetry with PSG as the gold standard | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine and Therapeutics, Prince of Wales Hospital, CUHK, Hong Kong, Hong Kong